CLINICAL TRIAL: NCT06175026
Title: Encouraging Healthy and Sustainable Dietary Substitutions: A Randomized Experiment With Emerging Adults
Brief Title: Encouraging Healthy and Sustainable Dietary Substitutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anna Grummon, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 71737; K01HL158608 (NIH)
Record Dates: First submitted 2023-11-30; First posted 2023-12-18 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Food Selection
Keywords: health; environment; sustainability; food choices; dietary substitutions; diet; emerging adults
MeSH Terms: conditions — Food Preferences | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Health messages (Experimental): Messages shown will be related to the health impacts of making certain dietary substitutions (replacing beef with chicken and vegetarian entrees; replacing juice with whole fruit; replacing dairy milk with non-dairy milk; replacing sugar-sweetened beverages with water).
  Interventions: Behavioral: Health messages
- Environment messages (Experimental): Messages shown will be related to the environmental impacts of making certain dietary substitutions (replacing beef with chicken and vegetarian entrees; replacing juice with whole fruit; replacing dairy milk with non-dairy milk; replacing sugar-sweetened beverages with water).
  Interventions: Behavioral: Environmental messages
- Health and environment messages (Experimental): Messages shown will be related to the health and environmental impacts of making certain dietary substitutions (replacing beef with chicken and vegetarian entrees; replacing juice with whole fruit; replacing dairy milk with non-dairy milk; replacing sugar-sweetened beverages with water).
  Interventions: Behavioral: Health and environmental messages
- Neutral messages (Active Comparator): Messages shown will be neutral and unrelated to the health or environmental impacts of making certain dietary substitutions (replacing beef with chicken and vegetarian entrees; replacing juice with whole fruit; replacing dairy milk with non-dairy milk; replacing sugar-sweetened beverages with water).
  Interventions: Behavioral: Neutral messages

INTERVENTIONS:
Behavioral: Health messages — Participants view messages about the health impacts of certain dietary substitutions.
  Arms: Health messages
Behavioral: Environmental messages — Participants view messages about the environmental impacts of certain dietary substitutions.
  Arms: Environment messages
Behavioral: Health and environmental messages — Participants view messages about the health and environmental impacts of certain dietary substitutions.
  Arms: Health and environment messages
Behavioral: Neutral messages — Participants view neutral messages unrelated to the health and environmental impacts of certain dietary substitutions.
  Arms: Neutral messages

SUMMARY:
The aim of this study is to examine emerging adults' responses to dietary substitution messages about health, the environment, or both health and the environment.

DETAILED DESCRIPTION:
This online study will examine emerging adults' responses to dietary substitution messages about 4 different topics. Participants will be randomized to 1 of 4 topic arms: 1) Control (neutral topic, not related to health or the environment); 2) Health topic; 3) Environment topic; 4) Health and Environment topic. Participants will view messages about each of 4 dietary substitutions: replacing red meat with chicken or vegetarian options; replacing dairy milk with non-dairy milk; replacing juice with whole fruit; and replacing sugar-sweetened beverages with water. For each dietary substitution, participants will view 2 messages about their assigned topic, with the 2 messages shown in random order. Participants will rate each message on perceived message effectiveness (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-25 years
* Reside in the United States
* Ability to complete a survey in English

Exclusion Criteria:

* Older than 25 years; younger than 18 years
* Reside outside of the United States
* Unable to complete a survey in English

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1753 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grummon, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Stanford School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will post de-identified data to a public repository.
Supporting Information: SAP, Analytic Code
Time Frame: Investigators will post de-identified participant data upon acceptance of any manuscripts associated with the data generated in this study. Investigators will also share the statistical analysis plan and analytic code used for the study. The analysis plan will be uploaded before enrolling participants. The analytic code will be posted upon publication of manuscripts associated with data generated in this study.
Access Criteria: The data, statistical analysis plan, and analytic code will be publicly available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Messages | Environment Messages | Health and Environment Messages | Neutral Messages
Started | 441 | 446 | 431 | 435
Completed | 441 | 446 | 431 | 435
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: While 1,753 participants were randomized, 21 were excluded from the analysis: consistent with the pre-registration, 18 participants were excluded because they did not complete the survey and 3 participants were excluded because their survey completion time was determined to be too fast (i.e., participants completed the survey in less than 1/3 of the median completion time). Therefore, 1,732 participants were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Messages | Environment Messages | Health and Environment Messages | Neutral Messages | Total
Number analyzed (Participants) | 437 | 441 | 424 | 430 | 1732
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 437 | 441 | 424 | 430 | 1732
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (2.2) | 22.0 (2.3) | 21.9 (2.2) | 21.7 (2.3) | 21.8 (2.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 226 | 226 | 207 | 215 | 874
  Gender: Male | 196 | 210 | 207 | 205 | 818
  Gender: Non-binary or another gender | 15 | 5 | 10 | 10 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 60 | 80 | 76 | 271
  Not Hispanic or Latino | 382 | 381 | 344 | 354 | 1461
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 5 | 7 | 11 | 29
  Asian | 17 | 9 | 17 | 9 | 52
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 3 | 1 | 6
  Black or African American | 55 | 50 | 58 | 56 | 219
  White | 319 | 332 | 302 | 315 | 1268
  More than one race | 28 | 30 | 20 | 23 | 101
  Unknown or Not Reported | 10 | 15 | 17 | 15 | 57
Region of Enrollment [Number; unit: participants]
  United States | 437 | 441 | 424 | 430 | 1732

OUTCOME MEASURES:

1. Primary Outcome: Perceived Message Effectiveness
Description: Participants will rate each message on perceived message effectiveness (PME) for encouraging participants to make the target dietary substitution. PME will be assessed with 4 items [the text shown in brackets will be tailored to each substitution]:
  1. How much does this message discourage you from wanting to [eat beef and pork / drink juice / drink cow's milk / drink sugary drinks]?
  2. How much does this message make [eating beef and pork, etc.] seem unpleasant to you?
  3. How much does this message make you concerned about the effects of [eating beef and pork, etc.]?
  4. How much does this message make you want to [eat chicken or vegetarian options instead of beef and pork, etc.]?
  The response options for each item are: 1=Not at all, 2=Very little, 3=Somewhat, 4=Quite a bit, 5=A great deal.
  Investigators will average responses to these 4 items to create a perceived message effectiveness score. Higher scores indicated higher perceived message effectiveness.
Time Frame: Survey questions administered after participant viewed each message; overall survey took up to 20 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Messages | Environment Messages | Health and Environment Messages | Neutral Messages
Number analyzed (Participants) | 437 | 441 | 424 | 430
score on a scale | 2.94 (.95) | 2.83 (1.01) | 2.98 (.93) | 1.69 (.98)
Statistical Analysis 1: Comparison: Health Messages vs Neutral Messages; The null hypothesis was that the health messages would not elicit different levels of perceived message effectiveness compared to the neutral messages; Test type: Superiority; p < 0.001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [1.13 to 1.37], Standard Error of Mean .062
Statistical Analysis 2: Comparison: Environment Messages vs Neutral Messages; The null hypothesis was that the environment messages would not elicit different perceived message effectiveness than the control messages; Test type: Superiority; p < .001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. The a prior threshold for statistical significance was 0.05; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [1.03 to 1.26], Standard Error of Mean .062
Statistical Analysis 3: Comparison: Health and Environment Messages vs Neutral Messages; The null hypothesis was that the health and environment messages would not elicit different perceived message effectiveness than the control messages; Test type: Superiority; p < 0.001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons. The a prior threshold for statistical significance was 0.05; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [1.17 to 1.41], Standard Error of Mean .062
Statistical Analysis 4: Comparison: Health Messages vs Environment Messages; Test type: Superiority; p = .1892, Mixed Models Analysis — This p-value was adjusted for multiple comparisons (considering 3 tests among intervention arms) using the Bonferroni Holm method; Mean Difference (Final Values) = .10, 95% CI 2-sided [-0.018 to .223], Standard Error of Mean 0.062
Statistical Analysis 5: Comparison: Health Messages vs Health and Environment Messages; Test type: Superiority; p = .47, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 4]; Mean Difference (Final Values) = -.045, 95% CI 2-sided [-.17 to .08], Standard Error of Mean 0.62
Statistical Analysis 6: Comparison: Environment Messages vs Health and Environment Messages; Test type: Superiority; p = .051, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 4]; Mean Difference (Final Values) = -.15, 95% CI 2-sided [-.27 to -.03], Standard Error of Mean .062

ADVERSE EVENTS:
Time Frame: From the time of signing the Informed consent through study task completion, a total of approximately 20 minutes.
Arm/Group | Health Messages | Environment Messages | Health and Environment Messages | Neutral Messages
All-Cause Mortality (participants affected / at risk) | 0/437 | 0/441 | 0/424 | 0/430
Serious Adverse Events (participants affected / at risk) | 0/437 | 0/441 | 0/424 | 0/430
Other Adverse Events (participants affected / at risk) | 0/437 | 0/441 | 0/424 | 0/430

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT06175026/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT06175026/ICF_001.pdf